CLINICAL TRIAL: NCT03668158
Title: Multi-center Study on Therapy-oriented Molecular Subtyping of Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Xiao Xu, Clinical Professor, Zhejiang University
Other Study IDs: ZJHZXU2017
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- recurrent HCC: recurrent HCC after LT
- non-recurrent HCC: non- recurrent HCC after LT

SUMMARY:
The purpose of this study is to establish molecular subtyping of HCC.

DETAILED DESCRIPTION:
Hepatocellular carcinoma is one of the most common malignant tumors in the world with high incidence and mortality. Liver transplantation is the most effective treatment for HCC and is in high demand in China. However, recurrence of HCC among liver transplantation recipients is still a great challenge and threat to the survival of recipients. So it is of great significance to establish molecular subtyping of HCC and achieve precise selection of recipients. Based on large scales of samples, the investigator's study aims to establish multi-omics characteristic profiles of liver transplantation for HCC in integration of apparent biological characteristics, clinical management and prognostic information by utilizing genomics, transcriptomics and proteomics, etc. This study will contribute to the therapy-oriented molecular subtyping of HCC.

ELIGIBILITY:
Inclusion Criteria:

Liver transplantation due to HCC within Hangzhou criteria

Exclusion Criteria:

Liver transplantation due to HCC beyond Hangzhou criteria Liver transplantation due to other disease except HCC Multiple organ transplantation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalization patient
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-11-20 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
recurrence rate | 2 years